CLINICAL TRIAL: NCT03516981
Title: A Phase 2 Precision Oncology Study of Biomarker-Directed, Pembrolizumab-(MK-3475, SCH 900475) Based Combination Therapy for Advanced Non-Small Cell Lung Cancer (KEYNOTE-495; KeyImPaCT)
Brief Title: A Study of Biomarker-Directed, Pembrolizumab (MK-3475) Based Combination Therapy for Advanced Non-Small Cell Lung Cancer (MK-3475-495/KEYNOTE-495)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-495; MK-3475-495 (Other: MSD Protocol Number); 194621 (Registry Identifier: Japic-CTI); KEYNOTE-495 (Other: MSD); 2022-500990-16-00 (Registry Identifier: EU CT Number); 2017-003134-85 (EudraCT Number)
Record Dates: First submitted 2018-04-27; First posted 2018-05-07 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Advanced Non-Small Cell Lung Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- GEP low TMB low: Pembrolizumab + Quavonlimab (Experimental): Participants receive pembrolizumab 200 mg Q3W plus quavonlimab at the Recommended Phase 2 Dose ([RP2D], dose and schedule based on study NCT03179436) until disease progression, or until the participant has received 35 administrations of pembrolizumab (approximately 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Quavonlimab
- GEP low TMB low: Pembrolizumab + Favezelimab (Experimental): Participants receive pembrolizumab 200 mg Q3W plus favezelimab 200 mg or 800 mg Q3W until disease progression, or until the participant has received 35 administrations of pembrolizumab (approximately 2 years).
  Interventions: Biological: Pembrolizumab; Biological: Favezelimab
- GEP low TMB low: Pembrolizumab + Lenvatinib (Experimental): Participants receive pembrolizumab 200 mg Q3W plus lenvatinib 20 mg once daily until disease progression, or until the participant has received 35 administrations of pembrolizumab (approximately 2 years). Participants completing 35 infusions of pembrolizumab may continue with lenvatinib alone until disease progression or toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib
- GEP low TMB hi: Pembrolizumab + Quavonlimab (Experimental): Participants receive pembrolizumab 200 mg Q3W plus quavonlimab at the RP2D (dose and schedule based on study NCT03179436) until disease progression, or until the participant has received 35 administrations of pembrolizumab (approximately 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Quavonlimab
- GEP low TMB hi: Pembrolizumab + Favezelimab (Experimental): Participants receive pembrolizumab 200 mg Q3W plus favezelimab 200 mg or 800 mg Q3W until disease progression, or until the participant has received 35 administrations of pembrolizumab (approximately 2 years).
  Interventions: Biological: Pembrolizumab; Biological: Favezelimab
- GEP low TMB hi: Pembrolizumab + Lenvatinib (Experimental): Participants receive pembrolizumab 200 mg Q3W plus lenvatinib 20 mg once daily until disease progression, or until the participant has received 35 administrations of pembrolizumab (approximately 2 years). Participants completing 35 infusions of pembrolizumab may continue with lenvatinib alone until disease progression or toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib
- GEP hi TMB low: Pembrolizumab + Quavonlimab (Experimental): Participants receive pembrolizumab 200 mg Q3W plus quavonlimab at the RP2D (dose and schedule based on study NCT03179436) until disease progression, or until the participant has received 35 administrations of pembrolizumab (approximately 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Quavonlimab
- GEP hi TMB low: Pembrolizumab + Favezelimab (Experimental): Participants receive pembrolizumab 200 mg Q3W plus favezelimab 200 mg or 800 mg Q3W until disease progression, or until the participant has received 35 administrations of pembrolizumab (approximately 2 years).
  Interventions: Biological: Pembrolizumab; Biological: Favezelimab
- GEP hi TMB low: Pembrolizumab + Lenvatinib (Experimental): Participants receive pembrolizumab 200 mg Q3W plus lenvatinib 20 mg once daily until disease progression, or until the participant has received 35 administrations of pembrolizumab (approximately 2 years). Participants completing 35 infusions of pembrolizumab may continue with lenvatinib alone until disease progression or toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib
- GEP hi TMB hi: Pembrolizumab + Quavonlimab (Experimental): Participants receive pembrolizumab 200 mg Q3W plus quavonlimab at the RP2D (dose and schedule based on study NCT03179436) until disease progression, or until the participant has received 35 administrations of pembrolizumab (approximately 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Quavonlimab
- GEP hi TMB hi: Pembrolizumab + Favezelimab (Experimental): Participants receive pembrolizumab 200 mg Q3W plus favezelimab 200 mg or 800 mg Q3W until disease progression, or until the participant has received 35 administrations of pembrolizumab (approximately 2 years).
  Interventions: Biological: Pembrolizumab; Biological: Favezelimab
- GEP hi TMB hi: Pembrolizumab + Lenvatinib (Experimental): Participants receive pembrolizumab 200 mg Q3W plus lenvatinib 20 mg once daily until disease progression, or until the participant has received 35 administrations of pembrolizumab (approximately 2 years). Participants completing 35 infusions of pembrolizumab may continue with lenvatinib alone until disease progression or toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg pembrolizumab solution for intravenous (IV) infusion administered Q3W
  Other Names: MK-3475
Biological: Favezelimab — 200 mg or 800 mg favezelimab solution for IV infusion administered Q3W
  Other Names: MK-4280
  Arms: GEP hi TMB hi: Pembrolizumab + Favezelimab; GEP hi TMB low: Pembrolizumab + Favezelimab; GEP low TMB hi: Pembrolizumab + Favezelimab; GEP low TMB low: Pembrolizumab + Favezelimab
Drug: Lenvatinib — 20 mg lenvatinib capsules administered orally once daily
  Other Names: MK-7902
  Arms: GEP hi TMB hi: Pembrolizumab + Lenvatinib; GEP hi TMB low: Pembrolizumab + Lenvatinib; GEP low TMB hi: Pembrolizumab + Lenvatinib; GEP low TMB low: Pembrolizumab + Lenvatinib
Drug: Quavonlimab — Quavonlimab solution for IV infusion administered at the RP2D (dose and schedule based on study NCT03179436)
  Other Names: MK-1308
  Arms: GEP hi TMB hi: Pembrolizumab + Quavonlimab; GEP hi TMB low: Pembrolizumab + Quavonlimab; GEP low TMB hi: Pembrolizumab + Quavonlimab; GEP low TMB low: Pembrolizumab + Quavonlimab

SUMMARY:
This study will investigate the utility of biomarker-based triage for study participants with advanced non-small cell lung cancer (NSCLC) without prior systemic therapy. Study participants within groups defined by a biomarker-based classifier (gene expression profile [GEP] and tumor mutational burden [TMB]) will be randomized to receive pembrolizumab in combination with quavonlimab (MK-1308), favezelimab (MK-4280), or lenvatinib. The primary hypotheses are as follows: In participants receiving pembrolizumab in combination with either quavonlimab, favezelimab, or lenvatinib, the Objective Response Rate (ORR) will be 1) greater than 5% among participants with low GEP and low TMB, 2) greater than 20% among participants with low GEP and high TMB, 3) greater than 20% among participants with high GEP and low TMB, and 4) greater than 45% among participants with high GEP and high TMB.

DETAILED DESCRIPTION:
After Amendment 5, participants can receive 800 mg of favezelimab every 3 weeks (Q3W)

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically- or cytologically-confirmed diagnosis of Stage IV (American Joint Committee on Cancer [AJCC] v 8) NSCLC and has not had prior systemic therapy for advanced disease
* Has confirmation that epidermal growth factor receptor- (EGFR-), anaplastic lymphoma kinase- (ALK-), c-ros oncogene 1- (ROS1-), or B isoform of rapidly accelerated fibrosarcoma- (B-Raf-) directed therapy is not indicated as primary therapy (documentation of absence of tumor activating EGFR mutations, B-Raf mutations, ALK gene rearrangements, and ROS1 gene rearrangements)
* Has measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology
* Male participants must agree to use contraception during the treatment period and for ≥120 days, after the last dose of study treatment and refrain from donating sperm during this period. Male participants with pregnant partners must agree to use a condom
* Female participants eligible to participate if not pregnant, not breastfeeding, and not a woman of childbearing potential (WOCBP) or is a WOCBP who agrees to follow contraceptive guidance during the treatment period and for ≥120 days after the last dose of study treatment
* Provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Has adequate organ function

Exclusion Criteria:

* Has significant cardiovascular impairment within 12 months of the first dose of study drug: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or cerebrovascular accident (CVA) stroke, or cardiac arrhythmia associated with hemodynamic instability, significant cardiovascular impairment, or a left ventricular ejection fraction (LVEF) below the institutional normal range as determined by multigated acquisition scan (MUGA) or echocardiogram
* Prolongation of QTc interval to >480 milliseconds (ms)
* Has symptomatic ascites or pleural effusion
* Has had an allogenic tissue/solid organ transplant
* WOCBP who has a positive urine pregnancy test within 24 hours before the first dose of study treatment
* Has not recovered adequately from any toxicity and/or complications from major surgery prior to starting therapy, or has had major surgery within 3 weeks prior to first dose of study intervention
* Has preexisting ≥Grade 3 gastrointestinal or non-gastrointestinal fistula, gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib
* Radiographic evidence of major blood vessel invasion/infiltration
* Clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study drug
* Has received prior systemic chemotherapy treatment for metastatic/recurrent NSCLC
* Has current NSCLC disease that can be treated with curative intent with surgical resection, localized radiotherapy, or chemoradiation
* Is expected to require any other form of systemic or localized antineoplastic therapy while on study (including maintenance therapy with another agent for NSCLC, radiation therapy, and/or surgical resection)
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T cell receptor
* Has received previous treatment with another agent targeting the Lymphocyte-activation gene 3 (LAG-3) receptor
* Has received previous treatment with another agent targeting vascular endothelial growth factor (VEGF) or the VEGF receptor
* Has received prior anticancer therapy including investigational agents within 4 weeks prior to randomization
* Has received prior radiotherapy within 2 weeks of start of study treatment or received lung radiation therapy of >30 Gy within 6 months prior to the first dose of study intervention
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study treatment
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab, favezelimab, or lenvatinib and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs)
* Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection
* Has a known history of active tuberculosis (TB; Bacillus tuberculosis)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days (females and males) after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) | Up to ~2 years
  ORR was defined as the percentage of participants who have a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: At least a 30% decrease in the sum of diameters [SOD] of target lesions, taking as reference the baseline sum diameters) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) as assessed by local site.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) per RECIST 1.1 | Up to ~2 years
  PFS is defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to RECIST 1.1 as assessed by local site.
Overall Survival (OS) | Up to ~2 years
  OS is defined as the time from randomization to death due to any cause.
Number of Participants Experiencing Adverse Events (AEs) | Up to ~2 years
  An AE is any untoward medical occurrence in participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants in each treatment arm experiencing an AE will be reported.
Number of Participants Discontinuing Study Drug Due to AEs | Up to ~2 years
  An AE is any untoward medical occurrence in participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants in each treatment arm that discontinued study drug due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (81):
- United States (19):
  - Arizona Oncology Associates, PC- HAL ( Site 8001), Tempe, Arizona
  - University of California Davis Comprehensive Cancer Center ( Site 0137), Sacramento, California
  - University of California San Francisco ( Site 0111), San Francisco, California
  - UCLA Hematology/Oncology -Santa Monica ( Site 0108), Santa Monica, California
  - Yale University School of Medicine ( Site 0100), New Haven, Connecticut
  - Mayo Clinic Florida ( Site 0115), Jacksonville, Florida
  - University of Maryland ( Site 0136), Baltimore, Maryland
  - Mayo Clinic Rochester - St. Mary's Hospital ( Site 0117), Rochester, Minnesota
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0112), Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center ( Site 0113), New York, New York
  - Weill Cornell Medical College ( Site 0138), New York, New York
  - Oncology Hematology Care ( Site 8005), Cincinnati, Ohio
  - University of Pennsylvania ( Site 0132), Philadelphia, Pennsylvania
  - UPMC Cancer Center/Hillman Cancer Center ( Site 0104), Pittsburgh, Pennsylvania
  - Texas Oncology-Memorial City ( Site 8006), Houston, Texas
  - Texas Oncology-Tyler ( Site 8003), Tyler, Texas
  - Emily Couric Clinical Cancer Center ( Site 0134), Charlottesville, Virginia
  - Northwest Cancer Specialists, P.C. ( Site 8000), Vancouver, Washington
  - University of Wisconsin- Madison Carbone Cancer Center ( Site 0130), Madison, Wisconsin
- Australia (3):
  - Blacktown Hospital Western Sydney Local Health District ( Site 0200), Blacktown, New South Wales
  - Gallipoli Medical Research Foundation ( Site 0202), Brisbane, Queensland
  - Fiona Stanley Hospital ( Site 0201), Murdoch, Western Australia
- Canada (6):
  - The Ottawa Hospital ( Site 0306), Ottawa, Ontario
  - Sunnybrook Health Science Centre ( Site 0304), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0309), Toronto, Ontario
  - CIUSSS du Saguenay-Lac-St-Jean ( Site 0305), Chicoutimi, Quebec
  - Jewish General Hospital ( Site 0307), Montreal, Quebec
  - CIUSSS Ouest de l Ile - St-Mary s Hospital ( Site 0310), Montreal, Quebec
- Hong Kong (2):
  - Prince of Wales Hospital ( Site 1801), Hong Kong
  - Queen Mary Hospital ( Site 1800), Hong Kong
- Ireland (2):
  - St James Hospital ( Site 2200), Dublin
  - Mid Western Cancer Centre ( Site 2201), Limerick
- Italy (8):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori ( Site 0702), Meldola, Emilia-Romagna
  - Istituto Clinico Humanitas Research Hospital ( Site 0700), Rozzano, Lombardy
  - AOU San Luigi Gonzaga di Orbassano ( Site 0707), Orbassano, Torino
  - AULSS21 Regione Veneto Ospedale Mater Salutis - Legnago ( Site 0701), Legnago, Verona
  - Azienda Ospedaliera Papardo ( Site 0706), Messina
  - Seconda Universita degli Studi di Napoli ( Site 0704), Napoli
  - Fondazione Policlinico Universitario A. Gemelli ( Site 0703), Roma
  - Azienda Ospedaliera Universitaria Senese ( Site 0705), Siena
- Japan (2):
  - National Cancer Center Hospital ( Site 2001), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 2000), Tokyo
- Poland (3):
  - MED-POLONIA Sp. z o.o. ( Site 0907), Poznan, Greater Poland Voivodeship
  - Dolnoslaskie Centrum Onkologii. ( Site 0993), Wroclaw, Lower Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
- Russia (7):
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan ( Site 1003), Ufa, Baskortostan, Respublika
  - The Loginov Moscow Clinical Scientific Center ( Site 1008), Moscow, Moscow
  - N.N. Blokhin NMRCO ( Site 1000), Moscow, Moscow
  - Budgetary Healthcare Institution of Omsk Region Clinical Oncology Dispensary-Chemotherapy #1 ( Site, Omsk, Omsk Oblast
  - SBHI Leningrad Regional Clinical Hospital ( Site 1001), Saint Petersburg, Sankt-Peterburg
  - St Petersburg City Clinical Oncology Dispensary ( Site 1002), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 1005), Kazan', Tatarstan, Respublika
- Singapore (2):
  - National Cancer Centre Singapore ( Site 1900), Singapore, Central Singapore
  - National University Hospital ( Site 1901), Singapore, South West
- South Africa (7):
  - MPOC ( Site 2310), Groenkloof Pretoria, Gauteng
  - Wits Clinical Research ( Site 2313), Parktown-Johannesburg, Gauteng
  - Univ. Pretoria and Steve Biko Academic Hospitals ( Site 2315), Pretoria, Gauteng
  - Sandton Oncology Medical Group PTY LTD ( Site 2316), Sandton, Gauteng
  - Vaal Triangle Oncology Centre ( Site 2314), Vereeniging, Gauteng
  - Umhlanga Oncolgy Center ( Site 2311), Umhlanga, KwaZulu-Natal
  - Cape Town Oncology Trials Pty Ltd ( Site 2312), Kraaifontein, Western Cape
- South Korea (5):
  - Seoul National University Bundang Hospital ( Site 0803), Seongnam-si, Kyonggi-do
  - Asan Medical Center ( Site 0801), Songpa-gu, Seoul
  - Seoul National University Hospital ( Site 0800), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0802), Seoul
  - Samsung Medical Center ( Site 0805), Seoul
- Spain (3):
  - Hospital General Universitari Vall d Hebron ( Site 1100), Barcelona
  - Hospital Universitario Ramon y Cajal ( Site 1101), Madrid
  - Hospital Universitario 12 de Octubre ( Site 1102), Madrid
- Switzerland (5):
  - Kantonsspital St. Gallen ( Site 2102), Saint Gallen, Canton of Aargau
  - Universitaetsspital Basel ( Site 2104), Basel, Canton of Basel-City
  - Hopitaux Universitaires de Geneve HUG ( Site 2106), Geneva, Canton of Geneva
  - Universitaetsspital Zuerich ( Site 2100), Zurich, Canton of Zurich
  - Kantonsspital Graubuenden ( Site 2103), Chur, Kanton Graubünden
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital ( Site 1203), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 1202), Tainan
  - National Taiwan University Hospital ( Site 1200), Taipei
  - Taipei Veterans General Hospital ( Site 1204), Taipei
- United Kingdom (3):
  - Cambridge University Hospitals NHS Trust ( Site 1306), Cambridge, Cambridgeshire
  - University College London Hospital NHS Foundation Trust ( Site 1308), London, London, City of
  - Derriford Hospital ( Site 1301), Plymouth

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Gutierrez M, Lam WS, Hellmann MD, Gubens MA, Aggarwal C, Tan DSW, Felip E, Chiu JWY, Lee JS, Yang JC, Garon EB, Finocchiaro G, Ahn MJ, Luft A, Landers GA, Basso A, Ma H, Kobie J, Palcza J, Cristescu R, Fong L, Snyder A, Yuan J, Herbst RS. Biomarker-directed, pembrolizumab-based combination therapy in non-small cell lung cancer: phase 2 KEYNOTE-495/KeyImPaCT trial interim results. Nat Med. 2023 Jul;29(7):1718-1727. doi: 10.1038/s41591-023-02385-6. Epub 2023 Jul 10. PMID 37429923
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26334&tenant=MT_MSD_9011